CLINICAL TRIAL: NCT03919201
Title: Impacts of 12 Weeks of Resistance Band Exercise Training on Body Composition, Aging-related Hormones, and Blood Pressure in Postmenopausal Women With Hypertension
Brief Title: 12 Weeks of Resistance Band Exercise Impacts on Adiposity, Hormones, and Blood Pressure in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Responsible Party: Principal Investigator, Won-mok son, Principal Investigator, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PusanNU-4
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Hypertension; Hormone Disturbance; Adiposity
Keywords: postmenopausal; exercise
MeSH Terms: conditions — Hypertension; Endocrine System Diseases; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: exercise intervention group, control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): No exercise intervention
  Interventions: Other: No exercise intervention group
- Resistance band exercise intervention (Experimental): Exercise intervention group (resistance band exercise training for 12 weeks, 5x per week, for 60 minutes per day).
  Interventions: Other: Resistance band exercise intervention

INTERVENTIONS:
Other: Resistance band exercise intervention — Resistance band exercise intervention (12 weeks, 5x per week, 60 minutes per day)
  Arms: Resistance band exercise intervention
Other: No exercise intervention group — Control group: no exercise intervention
  Arms: Control group

SUMMARY:
The purpose of this study was to examine the impacts of a 12-week resistance band exercise program on body composition, aging-related hormones, and blood pressure in postmenopausal women with stage 1 hypertension. Twenty postmenopausal women with hypertension participated in this study. Participants were randomly allocated into the resistance band training group (EX, n = 10) or the control group (CON, n = 10). The EX group performed a resistance band exercise training program at jump rope training program at 40-70% of their heart rate reserve (HRR) 5 days/week for 12 weeks (sessions 60 minutes in duration). The CON group did not participate in any exercise, dietary, or behavioral intervention. Body composition, aging-related hormones (growth hormone, insulin-like growth factor 1, dehydroepiandrosterone, and estradiol), and blood pressure were measured before and after the 12-weeks study.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal
* hypertensive
* sedentary (no regular exercise training or physical activity within previous year)

Exclusion Criteria:

* premenopausal
* renal, pulmonary, and/or heart disease
* regularly physically active

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postmenopausal women (cessation of menses for a minimum of 12 consecutive months)
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
estradiol | 12 weeks
  Estradiol levels were measured pre- and post-exercise in picograms per milliliter (pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Song-Young Park, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Son WM, Pekas EJ, Park SY. Twelve weeks of resistance band exercise training improves age-associated hormonal decline, blood pressure, and body composition in postmenopausal women with stage 1 hypertension: a randomized clinical trial. Menopause. 2020 Feb;27(2):199-207. doi: 10.1097/GME.0000000000001444. PMID 31663986